CLINICAL TRIAL: NCT05552833
Title: Pulmonary Adaptive Responses to HIIT in COPD
Acronym: COPDEX0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Associate Professor, Principal investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COPDEX0
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: High intensity interval training (HIIT); Lung growth; Diffusion capacity; Blood flow; Lung tissue mass; Oxygen extraction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 12 COPD will undergo the intervention in one arm and 12 healthy, age and BMI matched individuals will undergo the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients (Experimental): This arm will consist of only COPD patients.
  Interventions: Other: High intensity interval training
- Healthy controls (Experimental): This arm will consist of age and BMI matched healthy controls.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — Participants will undergo 12 weeks of supervised HIIT training (3 times per week). The HIIT protocol will consist of 4x4 min.

SUMMARY:
Patients with chronic obstructive lung disease (COPD) suffer from a progressive loss of lung function that leads to poor quality of life, and often invalidity and early death. Regular exercise can improve quality of life in these patients, but the health care system lack the underlying mechanism of exercise-induced improvement in COPD and it is widely thought not to have any effect on lung function. The aim of the present study is to investigate to which extent lung tissue mass and rest-to-exercise diffusion capacity changes differ in COPD patients compared to the healthy state. In order to design prospective clinical trials on the putative impact of high-intensity interval training (HIIT) investigating these parameters, and a secondary aim is to assess the feasibility of such a study in terms of patient inclusion, adherence and methodology.

DETAILED DESCRIPTION:
Patients with Chronic obstructive pulmonary disease (COPD) suffer from a progressive loss of lung function that leads to poor quality of life, and often invalidity and early death. Regular exercise is considered the most effective non-pharmacological intervention for improving quality of life in these patients. However, its use is halted by the lack of understanding of the mechanism of exercise-induced improvement in COPD, and is widely thought not to have any effect on lung function in the clinical setting. Exercise is thus mainly considered a way to alleviate symptoms, primarily by improving skeletal muscle function, but without the potential to reverse the disease. Therefore, relatively short and low-intensity exercise interventions are typically prescribed and are often not pursued in patients with the greatest symptom burden.

The reasoning for not prescribing exercise more widely in COPD is based on two assumptions: 1) new tissue cannot be formed in the adult lung, and 2) no consistent exercise training-induced changes in lung function have previously been documented.

However, de novo tissue formation has repeatedly been demonstrated in the adult lung, both in animals and humans, primarily in response to prolonged hypoxia and pneumonectomy. It has recently been reported that interval-based training counteracts the progressive loss of lung tissue in animal models of experimental COPD. The most likely stimulus is the mechanical strain, and if any measurable changes are to be induced by training, a high-intensity interval training (HIIT) scheme is preferable to be initiated in pulmonary rehabilitation.

On this basis, this study aim to conduct a prospective randomised trial, in which the impact of HIIT on lung weight (assessed by CT), rest-to-exercise diffusion capacity, 3-dimensional distribution of pulmonary perfusion measured by single photon emission computed tomography (SPECT)-low dose CT are addressed. Indeed, the latter is an especially useful clinical tool for the pathophysiological classification of COPD patients, and rest-to-exercise SPECT has the potential as a diagnostic tool that 'pinpoints' the exact cause of dyspnoea in the individual COPD patient, but has not yet been validated for this purpose. While all the methods are established, there is a need for more information regarding COPD-associated changes in lung tissue mass ('lung weight') and rest-to-exercise pulmonary diffusion changes compared to the healthy state. An assessment of the feasibility of an extended HIIT-trial using these methods in COPD patients as well as estimates of the in-study changes in the resultant physiological estimates (for the purpose of sample size estimations) is warranted.

ELIGIBILITY:
Inclusion criteria -patients

* Men and women
* 45-80 years
* COPD (GOLD stage I to III)
* Forced expiratory volume in 1 sec (FEV1)/forced vital capacity ratio (FVC) < 0.8, FEV1 < 90% of predicted value
* Modified Medical Research Council score (mMRC 0 - 3)
* Resting arterial oxygenation > 90%
* Do not fulfil the physical activity recommendations by the Danish Health Authority

Inclusion criteria - controls

* Men and women
* 45-80 years
* Normal FEV1, FVC, FEV1/FVC, and single-breath diffusion capacity
* Same sex, age (± 3 years) and BMI (± 10%)
* Do not fulfil the physical activity recommendations by the Danish Health Authority (19)
* BMI 18-35

Exclusion criteria - patients

* Symptoms of ischaemic heart disease
* Known heart failure
* Previous severe or current COVID-19
* Unable to complete or understand HIIT training
* Claudication
* Symptoms of disease within 2 weeks prior to the study
* Participation in pulmonary rehabilitation within 6 months
* Known malignant disease
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Exclusion criteria - controls

* COPD
* Asthma
* Known ischaemic heart disease
* Known heart failure
* Previous severe or current COVID-19
* Unable to complete or understand HIIT training
* Symptoms of disease within 2 weeks prior to the study
* Known malignant disease
* Claudication
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Lung tissue mass | CT-scans at baseline and at 12 week follow up.
  Change in lung weight in COPD patients compared to matched controls using CT-scans.
Rest-to-exercise diffusion capacity | DLNO/CO measured at baseline and at 12 week follow up.
  Change in rest-to-exercise pulmonary diffusion capacity between COPD patients and matched healthy controls measured by DLNO/CO.

SECONDARY OUTCOMES:
Rest-to-exercise pulmonary perfusion ratio change | At baseline and at 12 week follow up
  Rest-to-exercise pulmonary perfusion ratio change in COPD patients compared to matched controls measured by single photon emission computed tomography (SPECT).
Rest-to-exercise leg blood flow change in COPD | At baseline and at 12 week follow up
  Rest-to-exercise leg blood flow change in COPD patients compared to matched controls measured by ultrasound doppler in a single leg knee extensor model.

OTHER OUTCOMES:
Rest-to-exercise cardiac output change | At baseline and at 12 week follow up
  Cardiac output measured by oxygen pulse.
VO2peak (and estimated VO2max) | At baseline and at 12 week follow up
  Incremental exercise test on bike ergometer with COSMED system using breath by breath analysis.
VO2 verification bout | At baseline and at 12 week follow up
  Confirmation of maximum oxygen consumption measured 20 minutes after intitial VO2 peak test at a 110 % of maximum workload.
The maximal workload (knee extension) | At baseline and at 12 week follow up.
  Incremental exercise test on one leg knee extensor chair.
Hand-grip strength | At baseline and at 12 week follow up.
  Measured with a dynamometer.
Body composition | At baseline and at 12 week follow up.
  total fat mass, lean body mass measured with dual energy x-ray absorption.
Lung function: FEV1 | At baseline and at 12 week follow up.
  Change in Forced expiratory volume in 1 second (FEV1) (ml)
Lung function: TLC | Measured during the 12 week intervention.
  Change in total lung capacity (TLC)(ml)
Lung function: FVC | Measured during the 12 week intervention.
  Change in forced vital capacity (FVC)(ml)
Lung function: RV | Measured during the 12 week intervention.
  Change in residual volume (RV) (ml)
Lung function: VA | Measured during the 12 week intervention.
  Change in alveolar volume (VA) (ml)
Lung function: DLCOc | Measured during the 12 week intervention.
  Single-breath diffusion capacity to carbon monoxide corrected for hemoglobin (ml/min/mmHg)
6-minute walking test | At baseline and at 12 week follow up.
  Distance transversed during 6 minutes of maximum effort walking.
Chronic obstructive pulmonary disease Assessment Test (CAT-score) | At baseline and at 12 week follow up.
  Health-related quality of life - COPD Assessment Test, (CAT) score. Higher values meaning a smaller burden of symptoms.
Oxygen extraction in lower limb musculature during small mass exercise | At baseline and at 12 week follow up.
  Calculated from paired arterial and venous blood gases obtained from intraarterial and venous catheters.
Intima media thickness in the carotid artery | At baseline and at 12 week follow up.
  Measured with ultrasound.
Exercise feasibility: exercise sessions attendance rate. | Measured during the 12 week intervention.
  Exercise attendance rate (%) defined as number of attended exercise sessions / by number of prescribed sessions x 100.
Exercise feasibility: Relative dose intensity (RDI) | Measured during the 12 week intervention.
  RDI (%) of exercise, defined as prescribed exercise dose / performed exercise dose x 100
Exercise feasibility: early exercise termination | Measured during the 12 week intervention.
  Incidence of early termination of attended exercise sessions, defined as termination of an exercise session before the prescribed exercises have been performed
Withdrawal rate | Measured during the 12 week intervention.
  Incidence of permanent discontinuations of the exercise intervention, defined as participants that withdraw entirely from the exercise intervention.
Exercise feasibility: Patient-reported symptomatic adverse events (paint, dizziness, nausea, fatigue, other) | Measured during the 12 week intervention.
  Changes in patient-reported symptomatic adverse events (pain, dyspnea, fatigue, cough, sore muscles)
Glucose | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of glucose
IL-1 | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of interleukin 1
IL-1RA | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of interleukin-1 receptor antagonist
TNF-alfa | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of tumor necrosis factor alfa
IL-6 | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of interleukin-6
IL-10 | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of interleukin 10
Adiponectin | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of adiponectin
IL-15 | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of interleukin 15
HS-CRP | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of high sensitive c-reactive protein
HDL | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of High density lipoprotein
LDL | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of low density lipoprotein
Insulin | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of insulin
Creatinine | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of creatinine
Leptin | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of leptin
Carbamide | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of carbamide
ALAT | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of alanine-aminotransferase
Leucocytes | At baseline and at 12 week follow up.
  Exercise induced changes in plasma levels of leucocytes

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Centre for Physical Activity Research (CFAS), Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
Can be retrieved upon request from primary investigator.